CLINICAL TRIAL: NCT05264064
Title: The Polish Version of the Alberta Infant Motor Scale: Cultural Adaptation and Validation
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Eliks, Principal Investigator, PhD student, Director of the project, Poznan University of Medical Sciences
Other Study IDs: 1034/19
Record Dates: First submitted 2022-02-10; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Infant Development
Keywords: Infant Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants aged 0-18 months: Healthy infants aged 0-18 months, divided into four age groups: 0-3 months, 4-7 months, 8-11 months, and older than 12 months
  Interventions: Other: The motor assessment to establish validation of the Polish version of the AIMS

INTERVENTIONS:
Other: The motor assessment to establish validation of the Polish version of the AIMS — The translation, cultural adaptation, and validation were conducted according to existing recommendations. The motor development of infants was assessed with the Polish scoresheet of the AlMS and the PDMS v.2. The examination was conducted by two peadiatric physiotherapists with a minimum 7 years of experience.The examination methodology was concordant with the recommendation of the authors of AIMS and PDMS-2.The intrarater reliability test included two assessments (with one-month interval) performed by one researcher (Rater A). For the second assessment, the videos of spontaneous motor performance of infants were recorded during the examination. The interrater reliability involved assessments by two researchers (Rater A, Rater B). The Gross Motor Scales of the PDMS v.2 was administered to estimate concurrent validity (participants at the age of 0-12 months).

SUMMARY:
The aim of the study was to derive a Polish version of the AIMS through its cultural adaptation and validation. This process was based on an analysis of intra- and interrater reliability, as well as concurrent validity, using PDMS-2.

DETAILED DESCRIPTION:
The monitoring infant motor development allows for detecting delays and disturbances, enabling, if necessary, early therapeutic interventions to prevent further structural and functional disorders. However, the developmental assessment should be performed using standardised tools, which need to undergo cultural adaptation adapted and validation. This process is necessary to ensure their reliability in countries, cultures, populations, and languages different than initially intended.

The Alberta Infant Motor Scale (AIMS) is a diagnostic tool for the developmental evaluation of infants from the time of birth, to the period of independent walking (0-18 months), based on the observation of spontaneous motor performance [9,10]. It is based on several assumptions of the neuromaturational model and the concepts of the dynamic systems development theory. The AIMS was created in the early 1990s by Piper and Darrah, validated and standardised on the Canadian population [9,10]. Moreover, a 2014 re-evaluation of the scale noted that the normative values in this population remained stable.

The intended uses of the AIMS comprise: 1) identification of infants with motor delay, 2) providing medical professionals and parents information on motor achievements of the infant (both currently developing activities and those not observed in the infant's repertoire), 3) measurement of motor performance over time, or before and after an intervention, 4) as a research tool for the estimation of rehabilitation program efficacy in infants with motor delays .

The scale has been used (as an outcome measure) in numerous studies in healthy infants and those affected by or at risk of developmental disorders.

So far, research on the reliability and validity of the AIMS has been performed in Japanese, Chinese, Brazilian, Spanish, Thai, Greek, Dutch, Flemish and Serbian sample groups. However, there has not yet been a study conducted in any Middle European population.

The aim of the study was to derive a Polish version of the AIMS through its cultural adaptation and validation. This process was based on an analysis of the intra- and interrater reliability, as well as concurrent validity, using PDMS-2.

ELIGIBILITY:
Inclusion Criteria:

* a gestational age between 37 and 42 weeks
* birth weight of ≥ 2500 g
* five-minute Apgar score ≥ 8.

Exclusion Criteria:

* a gestational age < 37 weeks,
* a birth weight < 2500 g,
* five-minute Apgar score < 8
* the presence of any neurological, orthopedic, genetic, metabolic, and sensory disorders.

Ages: 2 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study included 145 healthy infants aged 0-18 months, divided into four age groups: 0-3 months, 4-7 months, 8-11 months, and older than 12 months
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The reliability of the Polish version of the AIMS | 4 months
  The intrarater reliability test included two assessments (with one-month interval) of every participants with the Polish version AIMS performed by one researcher - a peadiatric physiotherapist (Rater A). For the second assessment, the videos of spontaneous motor performance of infants were recorded during the examination.
  The interrater reliability involved assessments of every participants by the Polish version of AIMS by two researchers - peadiatric physiotherapists (Rater A, Rater B).
  Intrarater and interrater reliability were examined via calculation of the intraclass correlation coefficient (ICC) and the 95% confidence interval (95%CI) of the ICC for the subscales, as well as total scores for the four studied age groups.

SECONDARY OUTCOMES:
The study of the concurrent validity of the Polish version of the AIMS | 12 months
  The concurrent validity was examined by the comparison the AIMS and the Gross Motor Scales of the Peabody Developmental Motor Scales v.2, which were administered to participants at the age of 0-12 months.
  Correlations between gross motor scales of PDMS-2 and AIMS were evaluated using the Spearman rank coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Eliks, Msc, Study Director — Poznan University of Medical Sciences, Department of Developmental Neurology
Locations (1):
- Poznan University of Medical Sciences, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mendonca B, Sargent B, Fetters L. Cross-cultural validity of standardized motor development screening and assessment tools: a systematic review. Dev Med Child Neurol. 2016 Dec;58(12):1213-1222. doi: 10.1111/dmcn.13263. Epub 2016 Oct 4. PMID 27699768
- [Result] Piper MC, Pinnell LE, Darrah J, Maguire T, Byrne PJ. Construction and validation of the Alberta Infant Motor Scale (AIMS). Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S46-50. PMID 1468050
- [Result] Saccani R, Valentini NC, Pereira KR. New Brazilian developmental curves and reference values for the Alberta infant motor scale. Infant Behav Dev. 2016 Nov;45(Pt A):38-46. doi: 10.1016/j.infbeh.2016.09.002. Epub 2016 Sep 13. PMID 27636655
- [Result] Fleuren KM, Smit LS, Stijnen T, Hartman A. New reference values for the Alberta Infant Motor Scale need to be established. Acta Paediatr. 2007 Mar;96(3):424-7. doi: 10.1111/j.1651-2227.2007.00111.x. PMID 17407470
- [Result] Wang H, Li H, Wang J, Jin H. Reliability and Concurrent Validity of a Chinese Version of the Alberta Infant Motor Scale Administered to High-Risk Infants in China. Biomed Res Int. 2018 Jun 13;2018:2197163. doi: 10.1155/2018/2197163. eCollection 2018. PMID 30009165
- [Result] Morales-Monforte E, Bagur-Calafat C, Suc-Lerin N, Fornaguera-Marti M, Cazorla-Sanchez E, Girabent-Farres M. The Spanish version of the Alberta Infant Motor Scale: Validity and reliability analysis. Dev Neurorehabil. 2017 Feb;20(2):76-82. doi: 10.3109/17518423.2015.1066461. Epub 2015 Aug 18. PMID 28125359
- [Result] Aimsamrarn P, Janyachareon T, Rattanathanthong K, Emasithi A, Siritaratiwat W. Cultural translation and adaptation of the Alberta Infant Motor Scale Thai version. Early Hum Dev. 2019 Mar;130:65-70. doi: 10.1016/j.earlhumdev.2019.01.018. Epub 2019 Jan 28. PMID 30703619
- [Derived] Eliks M, Anna S, Barbara S, Gajewska E. The standardization of the Polish version of the Alberta Infant Motor Scale. BMC Pediatr. 2023 May 12;23(1):236. doi: 10.1186/s12887-023-04055-5. PMID 37173690
- [Derived] Eliks M, Sowinska A, Gajewska E. The Polish Version of the Alberta Infant Motor Scale: Cultural Adaptation and Validation. Front Neurol. 2022 Jul 28;13:949720. doi: 10.3389/fneur.2022.949720. eCollection 2022. PMID 35968314